CLINICAL TRIAL: NCT03471793
Title: The Australian Colonic Large Sessile Lesion Endoscopic Resection Study
Acronym: ACE
Status: Recruiting | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Director of Interventional Endoscopy, Western Sydney Local Health District
Other Study IDs: HREC/16/WMEAD/383(4831)
Record Dates: First submitted 2018-03-13; First posted 2018-03-21 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colon Adenoma; Colon Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colonic polyp: Patients referred for EMR of a colonic polyp >20mm

SUMMARY:
A prospective, multicentre, observational study of all patients referred for endoscopic resection of sessile colorectal polyps sized ≥20 mm conducted with intention to treat analysis

DETAILED DESCRIPTION:
Colonoscopic polypectomy is well established as an effective way of reducing colorectal cancer mortality. The majority of polyps detected and removed at colonoscopy are adenomas <10mm in size without advanced histology. These lesions have a low risk of progression to malignancy and are relatively easily removed by standard snare polypectomy with low complication rates. Polyps that are sessile or flat and greater than 20mm in size are found in approximately 1% of all colonoscopies and are more difficult to manage. These lesions, known as large sessile lesions (LSL), have a high rate of advanced histology. Traditionally they have been managed by referral for open or laparoscopic surgery, which is definitive, but invasive, costly and associated with a significant mortality risk in patients with advanced age or comorbidities5. Endoscopic Mucosal Resection (EMR) has emerged in recent years as an alternative to surgery that is now becoming the standard of care. It is an outpatient procedure which is effective, safe and less costly than surgery when delivered at a tertiary referral centre6.

The Australian Colonic Endoscopic Mucosal Resection study (ACE), comprises two multicentre prospective observational studies which examined EMR of colonic LSL (Ethics approval No.s HREC JH/TG 2008/9/6.1(2858) and HREC/13/WMEAD/233 (3778)). The project now has an extensive dataset from leading colonic endoscopic resection centres in Australia on more than 2000 lesions resected over 4 years since September 2008.

These studies have been successful in addressing several aspects of the resection of LSL, resulting in several high profile papers in internationally recognised journals. The collection of this data has produced robust information on the efficacy of the procedure4, recurrence rates, bleeding complications and mortality and costs when compared to surgery. Single centre analysis of the ACE dataset at Westmead has also allowed insights into how to refine the procedure to improve outcomes. The target sign is now a recognised indication for the placement of clips to prevent perforation, CO2 insufflation for EMR has been shown to be superior to air insufflation and succinylated gelatin (Gelofusine®) has been shown to be superior to normal saline as a submucosal lifting agent. Assessment and management strategies for bleeding and deep mural injury or perforation have been derived from analysis of the data. Snare tip soft coagulation of the resection margin post-EMR has been shown to reduce recurrence in a randomised controlled trial. Several ACE study papers have been incorporated into review papers and international guidelines for the safe and effective performance of EMR.

There remain a number of unanswered questions regarding the endoscopic resection of large sessile lesions and a new study incorporating a greater number of endoscopy units around Australia will allow these to be addressed as well as answer questions on the clinical effectiveness of the technique. Enhancing the prediction of submucosal invasive cancer, advanced lesion classification, validation of the assessment of deep injury, treatment of lesion margins post resection to reduce recurrence, prevention and prophylaxis of bleeding, and subtype analyses of the different histological groups of colonic lesions will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for endoscopic resection of a large sessile colonic polyp or laterally spreading tumour ≥20mm in size.
* Able to give informed consent to involvement in the clinical study

Exclusion Criteria:

* Unable to provide informed consent for involvement

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for colonic EMR of a known sessile colonic polyp or laterally spreading lesion >20mm in size
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-02-24 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2037-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 6-60months
  Follow up colonoscopies as per standard of care for 6 - 60 months noting and treating any recurrence.

SECONDARY OUTCOMES:
Technical success for Endoscopic resection | 6-60 months
  To determine the safety, efficacy and predictors of success for Endoscopic Mucosal Resection of large sessile colorectal polyps.
Cancer prediction | peri-procedurally
  By properly assessing the lesion it is hoped that we will be able to provide the greater Gastroenterology community with a tool which can be used to properly identify benign and cancerous lesions to decrease the number of benign lesions being referred to surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia